CLINICAL TRIAL: NCT02041026
Title: Investigating the Effects of Probiotic Yoghurt on Reducing the Levels of Aflatoxin B1 Toxin Among the School Children in Eastern Kenya
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Technical University of Kenya (Other)
Collaborators: University of Western Ontario, Canada (Other)
Responsible Party: Principal Investigator, Nicholas Nduti, Food scientist, Technical University of Kenya
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: P446/08/2013
Record Dates: First submitted 2014-01-17; First posted 2014-01-20 (Estimated); Last update posted 2014-01-20 (Estimated); Status verified 2014-01

CONDITIONS: Aflatoxicosis
Keywords: probiotic; Yoghurt; NN20
MeSH Terms: conditions — Aflatoxin Poisoning

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- probiotic yoghurt (Experimental): the subject will be given 200ml of yogurt daily for 28 days
  Interventions: Dietary Supplement: probiotic yoghurt

INTERVENTIONS:
Dietary Supplement: probiotic yoghurt — The probiotic yoghurt will be prepared using lactobacillus NN20 isolated from Kimere (a traditional fermented food product) consumed in eastern part of kenya
  Other Names: NN20

SUMMARY:
We hypothesis that intake of probiotic yogurt reduces absorption of AFB1 in the gut and subsequently reduce AFM1 and aflatoxins adduct, the biomarker in human urine and blood respectively. We have demonstrated that yogurt made using weisella cibiria NN20 isolated from fermented dough made from pearl millet in eastern part of Kenya sequestered upto 42% of aflatoxin available in our invitro texts.

DETAILED DESCRIPTION:
In both the developed and developing world, humans are continuously exposed to a plethora of environmental toxins, both in nature and as the result of anthropomorphic activity. Aflatoxin B1, one such example, is one of the most toxic substances known to man, but it is all around us and can be found in our food, and especially cereals which form over 70% of Kenya staple food.

Limiting cereal intake is not always easy, as it is one of the most plentiful and nutritious food sources in Kenya and is the primary source of dietary energy for many societies in Kenya.

We have recently discovered a novel property of lactic acid bacteria in which aflatoxin B1, is sequestered and/or detoxified by the microbes causing reduction of toxin levels in their environment. We hypothesize that sequestration of toxins in the gastrointestinal tract by ingested probiotic bacteria will cause a reduction in host toxin uptake by carrying them out of the body in the feces preventing their passage from the gastrointestinal tract into the host. Our primary objective is to test our hypothesis that consumption of a probiotic yogurt will result in decreased levels of Aflatoxin B1 in a group of school-aged children. The secondary objective is to determine the baseline levels of aflatoxin B1 in a group of school-aged children in eastern Kenya. The tertiary objective is to establish the baseline gastrointestinal microbiota of these children and how consumption of a probiotic yogurt affects the microbiota.

A class of 60 pupils from Identified primary school, approximately 7 years old, will be randomized to two groups matching ages, sex and weight. They will receive a daily 100g serving of the probiotic yogurt and a portion of local milk in between the trial period. Before the first administration of the yogurt/milk, blood, urine and feces will be collected. After 30 days; biological specimens will again be collected to observe potential reductions in toxin levels.

ELIGIBILITY:
Inclusion Criteria:Participants will be recruited from an identified primary school and parental/ legal guardian consent will be required as well as assent from the child. The primary school has been identified with the help of Ministry of agriculture home economics extension officer. The criterion of selecting the primary school is accessibility from Embu ATC where yogurt will be produced and the area which is prone to aflatoxin B1. Children between the ages of 6 and 10 will be enrolled in the study.

-

Exclusion Criteria:Children would be excluded if they are already consuming fermented milk products or are lactose intolerant.

-

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2014-02; Primary Completion 2014-04 (Estimated); Study Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
Aflatoxin M1 in urine | 28 days
  urine samples will be collected from the subjects every morning before the first meal for a period of 28 days. Test of aflatoxin M1 the bio maker of aflatoxicosis will be carried in the samples.

SECONDARY OUTCOMES:
Albumin adduct in blood | 28 days
  baseline blood samples will be collected before intervetion and at the end of the study. test of albumin adduct in blood will be carried. this a bio maker of aflatoxicosis in blood

OTHER OUTCOMES:
microbiota in the stool | 28 days
  wewill analyze the intestinal microbiota of the children and to determine if consumption of a probiotic yogurt has a significant effect on the microbiota composition.

CONTACTS AND LOCATIONS:
Overall Officials: Gregor Reid, PhD, Study Director — Lawson health Research Institute- st Joseph hospital London Ontario; Nicholas Nduti, PhD expected, Principal Investigator — Technical University of Kenya
Locations (1):
- Embu, Embu, Embu County, Kenya

REFERENCES:
- See also: related infomation — http://globalnews.ca/news/996098/how-this-canadian-yogurt-is-detoxifying-the-worlds-food-supply/